CLINICAL TRIAL: NCT03633266
Title: Feasibility Study of Anti-VEGF Instead of Intraoperative PRP in Proliferative Diabetic Retinopathy
Brief Title: Anti-VEGF Instead of Intraoperative PRP in Proliferative Diabetic Retinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Xiangtian Zhou, professor, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10007
Record Dates: First submitted 2018-08-02; First posted 2018-08-16 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Anti-VEGF; Proliferative Diabetic Retinopathy; PRP; Vitrectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti-VEGF (Experimental): experimental group: vitreoretinal surgery combined with intraoperative anti-VEGF
  Interventions: Procedure: anti-VEGF
- PRP (Active Comparator): Control group: vitreoretinal surgery combined with intraoperative PRP
  Interventions: Procedure: PRP

INTERVENTIONS:
Procedure: anti-VEGF — vitreoretinal surgery combined with intraoperative anti-VEGF
  Arms: anti-VEGF
Procedure: PRP — vitreoretinal surgery combined with intraoperative PRP
  Arms: PRP

SUMMARY:
To evaluate the efficacy and safety of vitreoretinal surgery combined with anti-VEGF therapy in the replacement of intraoperative PRP in PDR therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old;
2. type 1 or type 2 diabetes.
3. proliferative diabetic retinopathy with vitreous hemorrhage, and conservative treatment of vitreous hemorrhage without obvious absorption for 1 month requires vitreoretinal surgery;
4. The postoperative refractive medium is clear and the pupil is large enough to obtain sufficient clear fundus

Exclusion Criteria:

1. Previously received panretinal photocoagulation or unfinished panretinal photocoagulation;
2. Pulling retinal detachment involving the macula or the presence of extensive fiber proliferation requires silicone oil filling;
3. anterior chamber neovascularization or neovascular glaucoma;
4. other vascular diseases such as retinal vein occlusion, arterial occlusion, etc;
5. received intraocular anti-VEGF therapy or triamcinolone acetonide treatment which are still in the treatment period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in best-corrected visual acuity (BCVA) | 3 years
  Assessed using the ETDRS protocol

SECONDARY OUTCOMES:
Mean change from baseline in visual field | 3 years
  Assessed on Humphery(30-2 and 60-4)
chang from baseline in sructure of retina | 3 years
  Assessed on Optical Coherence Tomography(OCT)
chang from baseline in retinal neovascularization | 3 years
  Assessed on Fundus Fluorescein Angiography(FFA)

CONTACTS AND LOCATIONS:
Overall Officials: Yong Wei, M.D, Principal Investigator — The Eye Hospital of Wenzhou Medical University